CLINICAL TRIAL: NCT05138562
Title: A Phase IIa, Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Proof of Concept Study to Evaluate the Efficacy and Safety of Orally Administered TU2670 in Subjects With Mod to Severe Endometriosis-Associated Pain
Brief Title: TUC3PII-01_TU2670 Phase IIa Clinical Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TiumBio Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TUC3PII-01
Record Dates: First submitted 2021-10-25; First posted 2021-12-01 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): 4 Placebo capsules
  Interventions: Drug: Placebo Comparator: Placebo
- TU2670 High Dose (Active Comparator): 320mg, QD
  Interventions: Drug: Active Comparator: TU2670 320mg
- TU2670 Medium Dose (Active Comparator): 240 mg, QD
  Interventions: Drug: Active Comparator: TU2670 240mg
- TU2670 Low Dose (Active Comparator): 120 mg, QD
  Interventions: Drug: Active Comparator: TU2670 120mg

INTERVENTIONS:
Drug: Placebo Comparator: Placebo — 4 x placebo capsules, QD
  Arms: Placebo
Drug: Active Comparator: TU2670 320mg — 320mg (80mg x 4), QD
  Arms: TU2670 High Dose
Drug: Active Comparator: TU2670 240mg — 240mg (80mg x 3 + placebo x 1), QD
  Arms: TU2670 Medium Dose
Drug: Active Comparator: TU2670 120mg — 120mg (80mg x 1 + 20mg x 2 + placebo x 1), QD
  Arms: TU2670 Low Dose

SUMMARY:
This Protocol for TU2670 is to investigate the efficacy, safety, pharmacokinetics (PK), and pharmacodynamics (PD) of multiple doses of TU2670 in subjects with moderate to severe endometriosis-associated pain.

DETAILED DESCRIPTION:
Treatment Groups and Duration:

Following a washout period of up to 12 weeks, subjects will enter a screening period of up to 12 weeks including an observation period consisting of a complete menstrual cycle.

Subjects will be randomly assigned in a 1:1:1:1 ratio to receive either 12 weeks of TU2670 320 mg QD, TU2670 240 mg QD, TU2670 120 mg QD, or matching placebo. TU2670 or a matching placebo will be administered in the clinic on Day 1. Subjects in the PK subset population will also receive the following additional doses in the clinic: Day 2 (after collection of the 24-hour PK sample); the dose on the day scheduled for subsequent serial PK sample collection (Week 4 or Week 5); and the next scheduled dose (after collection of the 24-hour PK sample). All other doses can be taken by the subject at home. Following the end of treatment, subjects will be followed up for safety for 12 weeks.

Statistical Methods:

All formal statistical tests will be done at the 5% 2-sided significance level. Point estimates will have 2 sided 95% confidence intervals (CIs) where applicable.

Where appropriate, variables will be summarized descriptively (frequency and percent will be summarized for categorical variables; n (number of available subjects), mean, standard deviation [SD], median, minimum, and maximum will be presented for continuous variables) by study visit and by treatment group.

Statistical summaries will be presented for the changes from baseline to each time point in efficacy endpoints that it is applicable.

ELIGIBILITY:
Inclusion Criteria:

* Independent Ethics Committee (IEC)-approved written informed consent/assent and privacy language as per national regulations must be voluntarily obtained from the subject.
* Premenopausal female subject, 18 to 45 years, inclusive
* Subject has moderate to severe endometriosis-related pain

Exclusion Criteria:

* Subject has used hormonal contraceptives or other drugs with effects on gynecological endocrinology within 12 weeks
* Subject has been nonresponsive to GnRH-agonist or antagonist therapy for the management of endometriosis.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
overall pelvic pain | 12 weeks
  Change from baseline to 12 weeks of treatment of the mean dysmenorrhea score (defined as mean overall pelvic pain score on menstrual bleeding days) as measured by the Numeric Rating Scale(minimum 0, maximum 10, higher score mean a worse outcome) over the past month.

SECONDARY OUTCOMES:
mean Numeric Rating Scale pain score | 12 weeks
  Change from baseline to 12 weeks of treatment of the mean Numeric Rating Scale pain score(minimum 0, maximum 10, higher score mean a worse outcome) for non-menstrual pelvic pain (mean Numeric Rating Scale pain score on non menstrual bleeding days)
mean overall pelvic pain Numeric Rating Scale pain score | 12 weeks
  Change from baseline to 12 weeks of treatment of the mean overall pelvic pain Numeric Rating Scale pain score (mean Numeric Rating Scale pain score(minimum 0, maximum 10, higher score mean a worse outcome) over all 28 days)
mean Numeric Rating Scale dyspareunia score | 12 weeks
  Change from baseline to 12 weeks of treatment of the mean Numeric Rating Scale((minimum 0, maximum 10, higher score mean a worse outcome) dyspareunia score
rescue medication | 12 weeks
  Change from baseline to 12 weeks of treatment of the use of protocol-defined rescue medication (ie, ibuprofen)
Time to increase of dose of rescue medication | 12 weeks
  Time to increase of dose of rescue medication from 0 week to 12 weeks
Time to decrease of dose of rescue medication | 12 weeks
  Time to decrease of dose of rescue medication from 0 week to 12 weeks
Modified Biberoglu and Behrman sign and symptom scores | 12 weeks
  Change from baseline to 12 weeks of treatment of the Modified Biberoglu and Behrman (mB&B) sign and symptom scores(minimum 0, maximum 3, higher score mean a worse outcome)
Patient Global Impression of Change | 12 weeks
  Patient Global Impression of Change (minimum 1, maximum 7, higher score mean a worse outcome) at 12 weeks of treatment
Endometriosis Health Profile-5 | 12 weeks
  Change from baseline to 12 weeks of treatment in the Endometriosis Health Profile-5 score(minimum 1(Never), maximum 5(Always), higher score mean a worse outcome)
36-Item Short Form Health Survey | 12 weeks
  Change from baseline to 12 weeks of treatment of the 36-Item Short Form Health Survey(Scoring meaning is different from the questions but usually lower score mean a worse outcome)
Work Productivity and Activity Impairment Questionnaire: General Health | 12 weeks
  Change from baseline to 12 weeks of treatment of the Work Productivity and Activity Impairment Questionnaire: General Health (Scoring meaning is different from the questions)

OTHER OUTCOMES:
Bone mineral density loss | 12 weeks
  Change from baseline to 12 weeks of treatment of the bone mineral density as assessed by dual-energy X-ray absorptiometry (DXA)

CONTACTS AND LOCATIONS:
Locations (40):
- Czechia (8):
  - University Hospital Hradec Kralove, Hradec Králové, Hradec Kralove
  - Kestr-gyn s.r.o., Gynekologicka ambulance, Náchod, Nachod
  - Fakultni Nemocnice Kralovske Vinohrady, Prague, Prague
  - OB/GYN, Prague, Praha 1
  - Vseobecna fakultni nemocnice v Praze, Dept. of Gynekologicko- porodnickaklinika 1.LF UK, Prague, Praha 2
  - University Hospital Brno, Brno
  - NEUMED gynekologicka ambulance, Olomouc
  - Nemocnice Na Bulovce, Prague
- Italy (8):
  - Università degli Studi di Cagliari - Policlinico Universitario Duilio Casula, Monserrato, Cagliari
  - Azienda ospedaliero-universitaria Senese, Siena, Tuscany
  - University of Florence, Florence
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico di Milano, Milan
  - AZIENDA Ospedaliero Univeritaria Di Modena, Modena
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
  - P.O. Sant'Anna, Torino
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Poland (11):
  - In Vivo sp. z o.o., Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Dolnośląskie Centrum Ginekologii, Wroclaw, Lower Silesian Voivodeship
  - Komed Centra Kliniczne, Lublin, Lublin Voivodeship
  - Hospital Pro-Familia, Rzeszów, Podkarpackie Voivodeship
  - Prywatna Klinika Położniczo-Ginekologiczna Sp. z o.o., Bialystok, Podlaskie Voivodeship
  - Centrum Medyczne Mikołowska, Katowice, Silesian Voivodeship
  - Examen sp z o.o., Skorzewo, Wielkopolska
  - Klinika Leczenia Niepłodności, Ginekologii i Położnictwa Bocian, Bialystok
  - Provita Sp. z o.o., Katowice
  - Klinika Leczenia Niepłodności, Ginekologii i Położnictwa Bocian, Fertility Clinic, Poznan
  - Gameta Hospital, Rzeszów, Łódź Voivodeship
- Russia (5):
  - Ural Research Institution of Maternity and Child Care of Russian Public Health Ministry, Yekaterinburg, Sverdlovsk Oblast
  - State Institution of Healthcare Moscow City Clinical Hospital # 13 of Moscow Department, Moscow
  - FSHI Clinical Hospital #85 of FMBA, Moscow
  - Moscow State University of Medicine and Dentistry, Moscow
  - SBIH Leningrad Regional Clinical Hospital, Saint Petersburg
- Ukraine (8):
  - Ivano-Frankivsk National Medical University on the basis of the municipal non-profit enterprise Ivano-Frankivsk Regional Perinatal Center of the Regional Council, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Communal non-commercial enterprise Vinnytsia City Clinical Hospital "Center of Mother and the Child, Vinnytsia, Vinnitsia
  - Communal Nonprofit Enterprise Maternity Hospital#4 of Zaporizhzhya Municipal Council, Zaporizhzhya, Zaporizhzhia Oblast
  - State Scientific Institution Center for Innovative Medical Technologies of the National Academy of Sciences of Ukraine, Kiev
  - Kyiv city clinical hospital #9, Department of gynecology, Kyiv
  - Lviv city clinical hospital #4, Lviv
  - Danylo Halytskyy Lviv national medical university, Lviv
  - Private Small-Scale Enterprise Medical Centre Pulse, Vinnytsia